CLINICAL TRIAL: NCT00019786
Title: A Phase II Study of Isolated Hepatic Perfusion (IHP) With Melphalan for Metastatic Unresectable Cancers of the Liver
Brief Title: Isolated Hepatic Perfusion With Melphalan in Treating Patients With Primary Unresectable Liver Cancer or Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 990123; 99-C-0123; CDR0000067220; NCT00001820 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer; Islet Cell Tumor; Liver Cancer; Metastatic Cancer; Neuroendocrine Carcinoma
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent islet cell carcinoma; adult primary hepatocellular carcinoma; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases; adult primary cholangiocellular carcinoma; advanced adult primary liver cancer; recurrent childhood liver cancer; childhood hepatocellular carcinoma; stage III childhood liver cancer; stage IV childhood liver cancer; neuroendocrine carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma, Islet Cell; Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Neuroendocrine; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Islet Cell | interventions — Melphalan

INTERVENTIONS:
Drug: isolated perfusion
Drug: melphalan
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well isolated hepatic perfusion with melphalan works in treating patients with primary unresectable liver cancer or liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response rate, duration of response, and patterns of recurrence in patients with primary or metastatic, unresectable cancers of the liver after treatment with isolated hepatic perfusion with melphalan.
* Determine the disease-free and overall survival of patients treated with this regimen.

OUTLINE: Patients who are otherwise eligible undergo an exploratory laparotomy of the peritoneal cavity. Patients with peritoneal seeding, unresectable extrahepatic metastases, or unresectable pathologically-involved lymph nodes outside area of portahepatis do not receive treatment. Remaining patients receive isolated hepatic perfusion with melphalan. Liver perfusion proceeds for 1 hour.

Patients are followed at 6 weeks, every 3 months for 2 years, and then every 4 months until disease progression.

PROJECTED ACCRUAL: A maximum of 67 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven liver cancer meeting 1 of the following criteria:

  * Primary unresectable hepatocellular or cholangiocellular carcinoma
  * Metastatic cancer to the liver originating from one of the following:

    * Intraocular melanoma (closed to accrual as of 10/17/03)
    * Islet cell carcinoma
    * Adenocarcinoma of the colon or rectum limited to parenchyma of the liver

      * No evidence of other unresectable extrahepatic colorectal metastasis
  * Other neuroendocrine tumors, such as carcinoid tumors
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 27.0%
* WBC at least 2,500/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL (3.0 mg/dL for patients with Gilbert's syndrome)
* PT no greater than 2 seconds above upper limit of normal
* Elevated SGOT and SGPT allowed if not due to hepatitis
* No biopsy-proven cirrhosis or evidence of significant portal hypertension
* No prior or concurrent veno-occlusive disease
* Patients with positive hepatitis B or C surface antigen serology and chronic active hepatitis are eligible provided there is no evidence of cirrhosis

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Congestive heart failure allowed if LVEF ≥ 40%

Pulmonary:

* No chronic obstructive pulmonary disease or other chronic pulmonary disease with pulmonary function tests less than 50% predicted for age

Other:

* Weight greater than 30 kg
* Not pregnant or nursing
* Negative pregnancy test
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 month since prior anticancer biologic therapy and recovered

Chemotherapy:

* At least 1 month since prior anticancer chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 month since prior anticancer radiotherapy and recovered

Surgery:

* Not specified

Other:

* Prior intrahepatic arterial infusion therapy allowed
* No chronic use of anticoagulants
* No concurrent immunosuppressive therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 1999-08; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Response rate
Duration of response
Patterns of recurrence
Disease-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: H. Richard Alexander, MD, FACS, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Feldman AL, Libutti SK, Pingpank JF, Bartlett DL, Beresnev TH, Mavroukakis SM, Steinberg SM, Liewehr DJ, Kleiner DE, Alexander HR. Analysis of factors associated with outcome in patients with malignant peritoneal mesothelioma undergoing surgical debulking and intraperitoneal chemotherapy. J Clin Oncol. 2003 Dec 15;21(24):4560-7. doi: 10.1200/JCO.2003.04.150. PMID 14673042